CLINICAL TRIAL: NCT02860845
Title: Multicenter Pilot Study to Compare the Efficacy of a Combination of Vaginal Capsules With Acid Boric, L.Gasseri and L.Rhamnosus Versus the Reference Medication in Patients With Vaginal Candidiasis or Bacterial Vaginosis
Brief Title: Use of Boric Acid in Combination With Probiotics for the Treatment of Vaginal Infections
Acronym: DOBO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratorios Ordesa (Industry)
Collaborators: Clever Instruments S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOBO-01-16
Record Dates: First submitted 2016-07-19; First posted 2016-08-09 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Candidiasis; Vaginosis, Bacterial
MeSH Terms: conditions — Candidiasis; Vaginosis, Bacterial | interventions — Anti-Bacterial Agents; Clindamycin; Antifungal Agents; Clotrimazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Boric acid and probiotics (Experimental): Boric acid with L.gasseri and L.rhamnosus
  Interventions: Device: Boric acid and probiotics
- Antibiotic/Antifungal (Active Comparator): Antibiotic: Clindamicine Antifungal: Clotrimazol
  Interventions: Drug: Antibiotic (Clindamycin); Drug: Antifungal (Clotrimazole)

INTERVENTIONS:
Device: Boric acid and probiotics — Vaginal capsules administered once a day during 7 days.
  Arms: Boric acid and probiotics
Drug: Antibiotic (Clindamycin) — Vaginal capsules containing a reference antibiotic (when bacterial vaginosis is suspected) administered once a day during 3 days.
  Other Names: Clindamycin
  Arms: Antibiotic/Antifungal
Drug: Antifungal (Clotrimazole) — Vaginal capsules containing a reference anti-fungal (when candidiasis is suspected) administered once a day during 6 days.
  Other Names: Clotrimazole
  Arms: Antibiotic/Antifungal

SUMMARY:
The purpose of this study is to determine whether a formula of boric acid and probiotics for vaginal application is effective in the treatment of symptomatic episodes of vulvovaginitis in comparison to pharmacological reference controls (depending on the suspected diagnosis).

DETAILED DESCRIPTION:
Multicentre, Open, Prospective, Randomized, Controlled. Women with suspected vaginal infection will be randomized and distributed into two groups (control or boric acid + probiotics). Follow-up will last for three months and consists in 3 visits and a telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years and agreement to participate by signing the consent form.
* Women with clinical manifestations of acute infectious vulvovaginitis (burning, pruritus, erythema, oedema, and abnormal vaginal discharge).

Exclusion Criteria:

* Clinical findings compatible with Chlamydia trachomatis, Neisseria gonorrhoeae or Trichomonas vaginalis infection.
* Use of anti-fungal, antibiotic or probiotic medication within last 2 weeks prior to the study.
* Patients receiving other treatment (drug, probiotics or vitamin supplements) that can significantly interfere with study evaluations during the 3 months of follow-up.
* Pregnant or high risk for pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan A Tena, Dr., Principal Investigator — Ginemed Sevilla
Locations (1):
- Ginemed Sevilla, Seville, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Boric Acid and Probiotics | Antibiotic/Antifungal
Started | 24 | 24
Analyzed Patients | 22 | 23
Completed | 22 | 23
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Boric Acid and Probiotics | Antibiotic/Antifungal | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.36 (8.2) | 37.7 (6.1) | 36.83 (7.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non latino | 23 | 24 | 47
  Latino | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Spain | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change in the Presence of Vaginitis Clinical Symptoms Determined by Sobel Score.
Description: Semi-quantitative scale where itching, erythema, edema, stinging and abnormal vaginal discharge are scored from 0 to 3: absent (0), mild (1), moderate (2), severe (3). Worse result is 3 (severe)
Time Frame: Baseline and at 2 weeks after treatment finalization
Population: Subscore Sobel Score values at baseline and visit 1 (from 0 to 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Boric Acid and Probiotics Baseline; Boric Acid and Probiotics Visit 1: Boric acid with L.gasseri and L.rhamnosus
  Boric acid and probiotics: Vaginal capsules administered once a day during 7 days.
- Antibiotic/Antifungal Baseline; Antibiotic/Antifungal Visit 1: Antibiotic: Clindamicine Antifungal: Clotrimazol
  Antibiotic (Clindamycin): Vaginal capsules containing a reference antibiotic (when bacterial vaginosis is suspected) administered once a day during 3 days.
  Antifungal (Clotrimazole): Vaginal capsules containing a reference anti-fungal (when candidiasis is suspected) administered once a day during 6 days.
Arm/Group | Boric Acid and Probiotics Baseline | Antibiotic/Antifungal Baseline | Boric Acid and Probiotics Visit 1 | Antibiotic/Antifungal Visit 1
Number analyzed (Participants) | 24 | 24 | 22 | 23
score on a scale
  Stinging sobel score | 1.13 (0.85) | 1.21 (1.06) | 0.18 (0.50) | 0.22 (0.67)
  Itching Sobel Score | 1.63 (0.85) | 1.58 (1.02) | 0.41 (0.80) | 0.57 (0.95)
  Erythema Sobel Score | 0.92 (0.93) | 0.96 (1.12) | 0.14 (0.64) | 0.17 (0.65)
  Edema Sobel Score | 0.5 (0.78) | 0.42 (0.72) | 0.05 (0.21) | 0 (0.00)
  abnormal vaginal discharge | 1.67 (0.96) | 1.96 (1.08) | 0.23 (0.53) | 0.35 (0.83)

2. Secondary Outcome: Change in the Level of Lactobacillus in Vaginal Flora Determined by Vaginal Cultures.
Description: Lactobacillus spp count. in vaginal discharge at baseline and at visit 1, determined by vaginal cultures.
Time Frame: Baseline and 2 weeks after treatment finalization
Measure: Mean (Standard Deviation); unit: Count of Organism/counting chamber
Arm/Group | Boric Acid and Probiotics Baseline | Antibiotic/Antifungal Baseline | Boric Acid and Probiotics Visit 1 | Antibiotic/Antifungal Visit 1
Number analyzed (Participants) | 24 | 24 | 22 | 23
Count of Organism/counting chamber | 51.59 (50.74) | 49.30 (59.77) | 81.82 (84.34) | 66.09 (77.27)

3. Secondary Outcome: Number of Participants With Recurrent Infections
Description: Descriptive of the proportion of patients with vulvovaginitis recurrence
Time Frame: At 3 months after recruitment
Measure: Count of Participants; unit: Participants
Arm/Group | Boric Acid and Probiotics | Antibiotic/Antifungal
Number analyzed (Participants) | 22 | 23
Participants
  No recurrence | 17 | 14
  Recurrence | 5 | 9

ADVERSE EVENTS:
Time Frame: From baseline to three months
Arm/Group | Boric Acid and Probiotics | Antibiotic/Antifungal
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT02860845/Prot_SAP_000.pdf